CLINICAL TRIAL: NCT01297881
Title: Belgian Pulmonary Function Study : the Belgian Thoracic Society
Brief Title: Belgian Pulmonary Function Study
Acronym: BPFS
Status: Completed | Type: Observational
Sponsor: Marc Decramer (Other)
Collaborators: Belgian Pulmonary Society (Unknown)
Responsible Party: Sponsor-Investigator, Marc Decramer, MD PhD, KU Leuven
Organization: KU Leuven (Other)
Other Study IDs: S52460
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Respiratory Symptoms
Keywords: Caucasian outpatients; undiagnosed respiratory symptoms; dyspnea; cough; sputum
MeSH Terms: conditions — Signs and Symptoms, Respiratory; Dyspnea; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Caucasian outpatients with respiratory symptoms: all consecutive new Caucasian outpatients with respiratory symptoms like dyspnoea, cough, sputum but without diagnosis who are being examined for the first time.

SUMMARY:
Pulmonary function tests including spirometry, lung volumes, measurements of resistance and diffusing capacity are essential in the diagnosis of several pulmonary diseases. These tests are an integral part of the diagnosis and treatment of lung diseases, but until now there is no clear evidence for the use of many of the pulmonary function tests because of a lack of adequate studies. The obscurity largely pertains to the conditions under which combinations of the various tests are indicated. Therefore the Belgian Thoracic Society, assembling all pulmonologists and the pneumology LOK/GLEM"s, will investigate this matter.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age between 18 and 75 years old
* New outpatients with respiratory symptoms as dyspnoea, cough, sputum, but without firm diagnosis
* Results of the tests are available and acceptable
* Standardized list of complaints
* Capability of patient for doing pulmonary function tests
* Seen by a Pneumologist
* Written informed consent

Exclusion Criteria:

* Patients with diagnosed respiratory disease
* Younger than 18 and older than 75 years old
* Recent heart attack
* Pneumothorax
* hemoptoic
* Suspicion of Tuberculosis
* Not capable to do pulmonary function tests

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caucasian outpatients with respiratory symptoms but without diagnosis
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
pulmonary function tests (spirometry, volumes, resistance and diffusing capacity in that order) on the preferential diagnosis. | end of study
  To determine the effect of stepwise addition of various pulmonary function tests (spirometry, volumes, resistance and diffusing capacity in that order) on the preferential diagnosis and its reflection of the gold standard (final diagnosis), a statistical score will be calculated based on 1/n differential diagnoses after every pulmonary function test. The score will contain corrections for a high number of differential diagnoses and a wrong preferential diagnosis and compared with Linear mixed model after logistic transformation.

SECONDARY OUTCOMES:
% correct preferential diagnoses | end of study
  To determine the effect of stepwise addition of various pulmonary function tests (spirometry, volumes, resistance and diffusing capacity in that order) on preferential diagnoses and their reflection of the gold standard (final diagnosis), the number and percentage of correct preferential diagnoses will be analysed after every pulmonary function test and compared by a generalized estimating equation model (GEE)
N differential diagnoses in the subgroup with correct preferential diagnosis | end of study
  To determine the effect of stepwise addition of various pulmonary function tests (spirometry, volumes, resistance and diffusing capacity in that order) on the number of differential diagnoses and their reflection of the gold standard (final diagnosis), the number of differential diagnoses in patients with correct preferential diagnosis will be analysed after each pulmonary function test and compared with Poisson GEE
subgroup analyses | end of study
  The primary endpoint (1/n differntial diagnoses) and 2 secondary endpoints (% correct preferential diagnoses, n differential diagnoses within correct preferential diagnosis) will be analysed in subgroups with final gold standard diagnosis of COPD, asthma, interstitial lung disease and " no pulmonary abnormality"
Sensitivity analysis | end of study
  Primary endpoint (1/n differntial diagnoses) and 2 secondary endpoints (% correct preferential diagnoses, n differential diagnoses within correct preferential diagnosis) and subgroup analyses (asthma, COPD, interstitial lung disease and no primary pulmonary abnormality) will be evaluated not only considering final diagnosis as standard but als correct side diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Marc MD Decramer, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Flanders, Belgium

REFERENCES:
- [Derived] Decramer M, Janssens W, Derom E, Joos G, Ninane V, Deman R, Van Renterghem D, Liistro G, Bogaerts K; Belgian Pulmonary Function Study Investigators. Contribution of four common pulmonary function tests to diagnosis of patients with respiratory symptoms: a prospective cohort study. Lancet Respir Med. 2013 Nov;1(9):705-13. doi: 10.1016/S2213-2600(13)70184-X. Epub 2013 Oct 4. PMID 24429274